CLINICAL TRIAL: NCT00419601
Title: Prospective Randomized, Double-blinded Clinical Trial on Remifentanyl for Analgesia and Sedation of Ventilated Neonates and Infants
Brief Title: Rapip Study: Clinical Trial on Remifentanyl for Analgesia and Sedation of Ventilated Neonates and Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Prof. Dr. Bernhard Roth, Clinic for Paediatrics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KKSK 251; ISRCTN06135415 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-05

CONDITIONS: Mechanical Ventilation
Keywords: ventilated newborns (≥ 36 SSW)and infants (≤60 days); of any medical condition
MeSH Terms: interventions — Remifentanil; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Fentanyl
  Interventions: Drug: Fentanyl
- 1 (Experimental): Remifentanyl
  Interventions: Drug: Remifentanyl

INTERVENTIONS:
Drug: Remifentanyl — Start dose:9 µg/kg/h Maximum dose: 30 µg/kg/h
  Arms: 1
Drug: Fentanyl — start dose: 3 µg/kg/h Maximum dose: 10 µg/kg/h
  Arms: 2

SUMMARY:
It shall be investigated whether ventilated neonates and infants with a remifentanyl based analgesia and sedation can be extubated faster after discontinuation of the opioid infusion compared to neonates and infants with a fentanyl based analgesia and sedation.

DETAILED DESCRIPTION:
"Newborns (≥ 36 weeks of gestation) and young infants (≤ 60 days) with need of mechanical ventilation receive next to midazolam either remifentanyl or fentanyl for analgesia and sedation. The study medication will be started not later than 12 hours after intubation and the maximum application time is 96 hours. The opioid infusion rate is started with either 9µg/kg/h remifentanyl or 3µg/kg/h fentanyl and will be adapted according to a clinical sedation score (Hartwig- and Comfort score). The maximum infusion rate is 30µg/kg/h remifentanyl or 10µg/kg/h fentanyl.

To judge the efficacy of both opioids, we will evaluate the sedation scores every 6 hours and measure the skin conductance during a painful procedure (tracheal suctioning). Next to the adverse events we document different vital parameters like heart rate, blood pressure or oxygen saturation every 6 hours to estimate the safety of both opioids.

The midazolam plasma level will be determined immediately before termination of the opioid and midazolam infusion when the child is clinically judged to be ready for extubation. The child will be extubated as soon as it reaches a certain level in the sedation score and exhibits stable spontaneous breathing.

After extubation we will look in both treatment groups for the possible development of hyperalgesia by investigating the cutaneous flexor reflex with von Frey hairs. The trial ends for each patient 48 hours after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Ventilated term newborns and infants ≤ 60 days
* Expected time of artificial ventilation between 12 and 96 hours

Exclusion Criteria:

* Neuromuscular diseases
* Drug abuse of the mother (exclusion criteria for newborns)
* Known hypersensitivity to Ultiva® or Fentanyl-Janssen®
* Missing informed consent of the parents
* Participation in another clinical trial during the last 4 weeks before start of this trial

Max Age: 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2006-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Duration of the artificial ventilation after discontinuation of the opioid infusion | at time of extubation (expected to be within 48 hours following discontinuation of the opioid infusion)
  Extubation time point after discontinuation of the opioid infusion. Start of opioid infusion at the latest 12 h after intubation. Maximum duration of the opioid infusion 96 h.

SECONDARY OUTCOMES:
Efficacy of a remifentanyl based analgesia and sedation of mechanically ventilated newborns and infants | during opioid infusion
  During the opioid infusion we perform a score based evaluation every 6 hours. Start of opioid infusion at the latest 12 h after intubation. Maximum duration of the opioid infusion 96 h.
Safety of a continuous application of remifentanyl | up to 30 days after extubation
Possible withdrawal symptoms on both treatment groups after extubation | up to 48 h after extubation
Discharge time from the PICU after discontinuation of the opioid infusion | at time of discharge from the PICU (average 2 d after start of study medication)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Roth, Prof., Principal Investigator — Clinic for Paediatrics, University of Cologne
Locations (1):
- Clinic for Paediatrics, University of Cologne Kerpener Str. 62, Cologne, Germany

REFERENCES:
- [Derived] Welzing L, Oberthuer A, Junghaenel S, Harnischmacher U, Stutzer H, Roth B. Remifentanil/midazolam versus fentanyl/midazolam for analgesia and sedation of mechanically ventilated neonates and young infants: a randomized controlled trial. Intensive Care Med. 2012 Jun;38(6):1017-24. doi: 10.1007/s00134-012-2532-1. Epub 2012 Mar 29. PMID 22456770